CLINICAL TRIAL: NCT02808468
Title: Developing a Brief Early Cognitive Intervention for PTSD and Alcohol Misuse
Brief Title: Brief Restructuring Intervention Following Trauma Exposure
Acronym: BRITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Michele Bedard-Gilligan, Assistant Professor, Medicine: Psychiatry, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00003232; 1R34AA022966-01A1 (NIH)
Record Dates: First submitted 2016-06-17; First posted 2016-06-21 (Estimated); Results first posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Posttraumatic Stress Disorder; Alcohol Use Disorders
Keywords: Sexual assault; Posttraumatic Stress Disorder; Alcohol use; Cognitive therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Alcoholism; Alcohol Drinking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Cognitive Intervention (Active Comparator): One in person session (90 minutes) of trauma focused cognitive therapy followed by 4 weekly coaching calls (20 minutes each) with the same study therapist
  Interventions: Behavioral: Brief Cognitive Therapy
- Assessment Only (No Intervention): Assessment session followed by weekly completion of assessment measures

INTERVENTIONS:
Behavioral: Brief Cognitive Therapy — Cognitive strategies to help achieve balanced thinking around sexual assault and alcohol use
  Arms: Brief Cognitive Intervention

SUMMARY:
The broad aim of this study is to develop and test a brief intervention that can be implemented in the immediate weeks following sexual assault to decrease likelihood of developing posttraumatic stress disorder (PTSD) or alcohol misuse. The first phase of the study will enroll 6 women to complete a brief, cognitive therapy protocol and provide feedback on the intervention (open trial). The second phase of the study will recruit 76 women to complete either the intervention (38 women) or assessment only (38 women) to test the effects of the intervention on both PTSD symptoms and alcohol use behavior as compared to natural recovery following assault.

DETAILED DESCRIPTION:
Following sexual assault a substantial number of victims will go on to develop posttraumatic stress disorder (PTSD) or alcohol use disorders (AUD), and development of these disorders is costly to both the victim and society as a whole. Intervening early, in the initial weeks following sexual assault, can provide victims with coping strategies that can decrease the likelihood of developing chronic symptoms. Cognitive approaches for treating symptoms of PTSD have strong empirical support with chronic presentation of symptoms. Less is known about effective strategies for intervening acutely following sexual assault. This project is designed to adapt existing empirically supported cognitive treatment principles for both PTSD and AUD symptoms to be delivered acutely (within 10 weeks of assault) in a brief one session format followed by 4 weekly coaching calls. The first 6 participants enrolled will receive the intervention and provide us with feedback on strengths and weaknesses of the protocol to help us improve it (Open Trial). In the next phase, the pilot testing phase, the study will enroll 38 women to complete the one session intervention followed by 4 once per week coaching calls. Participants will then be assessed again for symptoms of PTSD and alcohol use behavior at 3 month follow-up. This brief intervention group will be compared at the 3 month follow-up to a group of 38 women who receive weekly symptom monitoring only. Thus, this research aims to provide information on the efficacy of the intervention compared to the natural recovery process. This research is significant in its potential to use a very brief and easy to access treatment to decrease the development of chronic psychopathology in a high risk group of women.

ELIGIBILITY:
Inclusion Criteria:

* Identifies as female
* Age > 18 years
* 2-10 weeks post sexual assault
* PTSD symptoms related to recent sexual assault, specifically defined as a minimum of

  1 reexperiencing, 1 avoidance, 2 negative alterations in mood/cognition, or 2 hyperarousal symptoms
* Drinking more than 3 drinks on one occasion in the last month and at least two reported negative consequences of alcohol use
* Capacity to provide informed consent
* English fluency
* No planned absences that they would be unable to complete 5 weeks of assessments and coaching calls
* Access to a telephone.

Exclusion Criteria:

* Acutely suicidal with intent/plan
* Exhibit current psychosis
* Previous non-response to an adequate trial (8 or more sessions) of Cognitive Processing Therapy (CPT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Must identify as female
Enrollment: 57 (Actual)
Dates: Start 2015-03-01; Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele Bedard-Gilligan, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bedard-Gilligan MA, Stappenbeck CA, Ojalehto HJ, Dworkin ER, Cadigan JM, Simpson T, Kaysen DL. A pilot randomized controlled trial of cognitive restructuring for PTSD and alcohol misuse following recent sexual assault: Initial efficacy and feasibility. Behav Res Ther. 2025 Oct;193:104847. doi: 10.1016/j.brat.2025.104847. Epub 2025 Aug 28. PMID 40925075
- [Derived] O'Doherty L, Whelan M, Carter GJ, Brown K, Tarzia L, Hegarty K, Feder G, Brown SJ. Psychosocial interventions for survivors of rape and sexual assault experienced during adulthood. Cochrane Database Syst Rev. 2023 Oct 5;10(10):CD013456. doi: 10.1002/14651858.CD013456.pub2. PMID 37795783

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Brief Cognitive Intervention | Assessment Only
Started | 28 | 29
Completed | 21 | 27
Not Completed | 7 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brief Cognitive Intervention | Assessment Only | Total
Number analyzed (Participants) | 28 | 29 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.1 (4) | 22.1 (3.4) | 21.6 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 29 | 57
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 24 | 26 | 50
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 5 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 16 | 22 | 38
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28 | 29 | 57
PTSD Symptom Severity [Mean (Standard Deviation); unit: score on a scale] — The Posttraumatic Stress Disorder Symptom Scale- Interview Version (PSS-I) assesses severity of symptoms of posttraumatic stress disorder (PTSD) as defined by the Diagnostic and Statistical Manual of Mental Disorders, fifth edition (DSM-5) and is administered at baseline and 3 month follow up to assess change in PTSD symptoms. The range for the scale is 0-80 with higher scores representing more severe PTSD symptoms.
  score on a scale | 32.4 (8.4) | 33.2 (8.4) | 32.8 (8.3)
Timeline Followback Heavy Episodic Drinking Episodes [Mean (Standard Deviation); unit: episodes] — The Timeline Followback (TLFB) uses a calendar method with cued recall to assess frequency and quantity of alcoholic beverages consumed. Quantity of drinks reported per day is used to calculate episodes of heavy episodic drinking (4+ drinks per occasion) and those are counted to calculate the number of HED episodes in the past month. The minimum score possible is 0 for number of HED episodes in the past month and the maximum is 30 (count of days in past 30 days in which HED occurred). Higher numbers indicate more heavy episodic drinking episodes.
  episodes | 5.4 (4.4) | 5.8 (3.5) | 5.6 (3.9)
Alcohol use negative consequences [Mean (Standard Deviation); unit: score on a scale] — Total score of alcohol related negative consequences as reported on the self-report Drinking Inventory of Consequences (DrInC). The total range of scores is 0-135 and higher scores indicate more negative consequences of alcohol use. It is administered at baseline and 3-month follow-up to assess change in alcohol related consequences.
  score on a scale | 17.7 (24.3) | 19.8 (15.3) | 18.74 (20.1)

OUTCOME MEASURES:

1. Primary Outcome: Posttraumatic Stress Disorder Symptom Scale- Interview Version (PSS-I)
Description: The Posttraumatic Stress Disorder Symptom Scale- Interview Version (PSS-I) assesses severity of symptoms of posttraumatic stress disorder (PTSD) as defined by the Diagnostic and Statistical Manual of Mental Disorders, fifth edition (DSM-5) and is administered at baseline and 3 month follow up to assess change in PTSD symptoms. The range for the scale is 0-80 with higher scores representing more severe PTSD symptoms.
Time Frame: 12 weeks
Population: Analyzed data from all participants assigned to each condition regardless of completion or missing data (intent to treat).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brief Cognitive Intervention | Assessment Only
Number analyzed (Participants) | 28 | 29
score on a scale | 11.4 (7.0) | 22.1 (10.4)

2. Primary Outcome: Timeline Followback Heavy Episodic Drinking Episodes
Description: The Timeline Followback (TLFB) uses a calendar method with cued recall to assess frequency and quantity of alcoholic beverages consumed. Quantity of drinks are reported per day. Episodes of heavy episodic drinking (4+ drinks per occasion) are counted to calculate the number of HED episodes in the past month. The minimum score possible is 0 for number of HED episodes in the past month and the maximum is 30 (count of days in past 30 days in which HED occurred). Higher numbers indicate more heavy episodic drinking episodes.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: episodes
Arm/Group | Brief Cognitive Intervention | Assessment Only
Number analyzed (Participants) | 28 | 29
episodes | 2.2 (2.7) | 3.7 (3.7)

3. Secondary Outcome: Drinking Inventory of Consequences (DrInC)
Description: Total score of alcohol related negative consequences as reported on the self-report Drinking Inventory of Consequences (DrInC). The total range of scores is 0-135 and higher scores indicate more negative consequences of alcohol use. It is administered at baseline and 3-month follow-up to assess change in alcohol related consequences.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brief Cognitive Intervention | Assessment Only
Number analyzed (Participants) | 28 | 29
score on a scale | 7.4 (14.0) | 19.8 (15.3)

ADVERSE EVENTS:
Time Frame: 3 months
Description: Study followed definitions of adverse event and serious adverse event used in clinicaltrials.gov. Adverse event information was collected at 3-month follow-up interview.
Arm/Group | Brief Cognitive Intervention | Assessment Only
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/29
Other Adverse Events (participants affected / at risk) | 0/28 | 0/29

LIMITATIONS AND CAVEATS:
Recruitment was ended before reaching target enrollment due to slower than anticipated recruitment and the COVID-19 pandemic which necessitated pausing all in person research activities at our site. Funding expired during the pandemic and we were not able to resume recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2014-03-08): https://cdn.clinicaltrials.gov/large-docs/68/NCT02808468/Prot_SAP_000.pdf
  • Informed Consent Form (2017-05-02): https://cdn.clinicaltrials.gov/large-docs/68/NCT02808468/ICF_001.pdf